CLINICAL TRIAL: NCT06734234
Title: A Randomised, Double Blind, Placebo-controlled, Single Ascending Dose, Phase 1a/1b Multi-centre Study in Healthy Participants and Participants With Autosomal Dominant Polycystic Kidney Disease to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of GSK4771261
Brief Title: A Study to Evaluate the Safety, Tolerability, and Effects on Blood and Urine Markers of Single Ascending Dose of GSK4771261 in Healthy Participants and Participants With Autosomal Dominant Polycystic Kidney Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 221362; 2024-516095-15 (Other: EU CT Number)
Record Dates: First submitted 2024-12-11; First posted 2024-12-16 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Kidney Disease
Keywords: Phase 1; GSK4771261; Autosomal dominant polycystic kidney disease (ADPKD); Safety; Tolerability; Pharmacokinetics; Pharmacodynamics; Immunogenicity
MeSH Terms: conditions — Kidney Diseases; Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Intervention Model Description: This is sequential double-blind study.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (15):
- Part A: Cohort 1: Participants receiving GSK4771261 Dose level 1 (Experimental): Healthy participants will be randomized to receive GSK4771261 Dose level 1.
  Interventions: Drug: GSK4771261
- Part A: Cohort 2 : Participants receiving GSK4771261 Dose level 2 (Experimental): Healthy participants will be randomized to receive GSK4771261 Dose level 2.
  Interventions: Drug: GSK4771261
- Part A: Cohort 3: Participants receiving GSK4771261 Dose level 3 (Experimental): Healthy participants will be randomized to receive GSK4771261 Dose level 3.
  Interventions: Drug: GSK4771261
- Part A: Cohort 4: Participants receiving GSK4771261 Dose level 4 (Experimental): Healthy participants will be randomized to receive GSK4771261 Dose level 4.
  Interventions: Drug: GSK4771261
- Part A: Cohort 5: Participants receiving GSK4771261 Dose level 5 (Experimental): Healthy participants will be randomized to receive GSK4771261 Dose level 5.
  Interventions: Drug: GSK4771261
- Part A: Cohort 6: Participants receiving GSK4771261 Dose level 6 (Experimental): Healthy participants will be randomized to receive GSK4771261 Dose level 6.
  Interventions: Drug: GSK4771261
- Part A: Cohort 7 (optional): Participants receiving GSK4771261 Dose level 7 (Experimental): Healthy participants will be randomized to receive GSK4771261 Dose level 7 as the recommendation of Dose escalation committee (DEC).
  Interventions: Drug: GSK4771261
- Part A: Cohort 8 (optional): Participants receiving GSK4771261 Dose level 8 (Experimental): Healthy participants will be randomized to receive GSK4771261 Dose level 8, as per the recommendation from DEC.
  Interventions: Drug: GSK4771261
- Part B: Cohort 1: Participants receiving GSK4771261 Dose level 9 (Experimental): Participant with Autosomal dominant polycystic kidney disease (ADPKD) will be randomized to receive GSK4771261 Dose level 9.
  Interventions: Drug: GSK4771261
- Part B: Cohort 2: Participants receiving GSK4771261 Dose level 10 (Experimental): Participant with ADPKD will be randomized to receive GSK4771261 Dose level 10.
  Interventions: Drug: GSK4771261
- Part B: Cohort 3: Participants receiving GSK4771261 Dose level 11 (Experimental): Participant with ADPKD will be randomized to receive GSK4771261 Dose level11.
  Interventions: Drug: GSK4771261
- Part B: Cohort 4 (optional): Participants receiving GSK4771261 Dose level 12 (Experimental): Participant with ADPKD will be randomized to receive GSK4771261 Dose level 12 as the recommendation from DEC.
  Interventions: Drug: GSK4771261
- Part B: Cohort 5 (optional): Participants receiving GSK4771261 Dose level 13 (Experimental): Participant with ADPKD will be randomized to receive GSK4771261 Dose level 13, as per the recommendation from DEC.
  Interventions: Drug: GSK4771261
- Part A: Participants receiving Placebo matching GSK4771261 (Placebo Comparator): Participants will receive placebo matching GSK4771261
  Interventions: Drug: Placebo matching GSK4771261
- Part B: Participants receiving placebo matching GSK4771261 (Placebo Comparator): Participants will receive placebo matching GSK4771261
  Interventions: Drug: Placebo matching GSK4771261

INTERVENTIONS:
Drug: GSK4771261 — GSK4771261 will be administered.
  Arms: Part A: Cohort 1: Participants receiving GSK4771261 Dose level 1; Part A: Cohort 2 : Participants receiving GSK4771261 Dose level 2; Part A: Cohort 3: Participants receiving GSK4771261 Dose level 3; Part A: Cohort 4: Participants receiving GSK4771261 Dose level 4; Part A: Cohort 5: Participants receiving GSK4771261 Dose level 5; Part A: Cohort 6: Participants receiving GSK4771261 Dose level 6; Part A: Cohort 7 (optional): Participants receiving GSK4771261 Dose level 7; Part A: Cohort 8 (optional): Participants receiving GSK4771261 Dose level 8; Part B: Cohort 1: Participants receiving GSK4771261 Dose level 9; Part B: Cohort 2: Participants receiving GSK4771261 Dose level 10; Part B: Cohort 3: Participants receiving GSK4771261 Dose level 11; Part B: Cohort 4 (optional): Participants receiving GSK4771261 Dose level 12; Part B: Cohort 5 (optional): Participants receiving GSK4771261 Dose level 13
Drug: Placebo matching GSK4771261 — Placebo matching GSK4771261 will be administered.
  Arms: Part A: Participants receiving Placebo matching GSK4771261; Part B: Participants receiving placebo matching GSK4771261

SUMMARY:
This is a study where a new drug, called GSK4771261 is being tested. Neither the study doctors, study staff or participants will be aware of what treatment is being given. Part A is testing the new study treatment on healthy people. This is to see if it's safe, what it does to the body, and how the body's defense system responds to it. Part B is similar, but the study treatment will be given to people who have a kidney disease called autosomal dominant polycystic kidney disease (ADPKD).

ELIGIBILITY:
Inclusion Criteria:

For Part A

* Body weight greater than or equal to (>=) 45 kilograms (kg) and basal metabolic index (BMI) within the range 19.5 to 32 kilograms per square meters (kg/m^2), inclusive
* Capable of giving signed informed consent,
* Participants who are overtly healthy as determined by medical evaluation by the investigator or a medically qualified designee based on medical history, physical examination, laboratory tests, and cardiac monitoring
* Women must be of non-childbearing potential

For Part B (planned Cohorts 1-3 and optional cohorts 4-5):

* Body weight >=45 kg and BMI within the range 19.5 to 32 kg/m^2, inclusive.
* Capable of giving signed informed consent, Confirmed diagnosis of Autosomal dominant polycystic kidney disease (ADPKD) by either applicable guidelines and/or genetic and imaging screening assessments
* Participants diagnosed with ADPKD may have complications or comorbidities directly related to ADPKD but should be otherwise healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests clinical testing
* Confirmation of known ADPKD causal genetic mutation(s) at the Polycystic kidney disease (PKD)1 and/or PKD2 loci based on genetic testing at screening and/or existing genetic information collected during the participant's routine clinical care for ADPKD from a genetic testing provider that, in the judgement of the investigator, is clinically valid.
* Mayo imaging classification groups 1C, 1D or 1E as assessed using the information collected at screening
* Estimated glomerular filtration rate (eGFR) greater than or equal to (>=) 45 milliliters per minutes per 1.73 square meters (mL/min/1.73m^2) (based on the Chronic kidney disease- Epidemiology Collaboration [CKD-EPI 2021] eGFR equation) and is not anticipated by the participant's regular treating physician to have a sustained decline by greater than (>)10 percent (%) over the following 12 months
* Intolerant of tolvaptan treatment, unwilling to initiate tolvaptan treatment or ineligible for tolvaptan treatment for ADPKD
* A female participant is eligible to participate if she is not pregnant or breastfeeding and agrees to use birth control methods as discussed with the study doctor.
* Woman of childbearing potential (WOCBP) and Woman of non-childbearing potential (WONCBP) must have a negative highly sensitive pregnancy test prior to the Magnetic resonance imaging (MRI) scan being performed in the screening period of Part B
* A WOCBP and WONCBP must have a negative highly sensitive pregnancy test (urine or serum as required by local regulations) within 24 hours before the first dose of study intervention For Part B (additional inclusion criteria for optional cohorts 4-5 only)
* eGFR >=30 mL/min/1.73m^2 (based on the CKD-EPI 2021 eGFR equation) and, in the clinical judgement of the investigator, the participant:
* has been clinically stable for the 24 months before screening; and,
* is not anticipated by the participant's regular treating physician to have a sustained decline in kidney function by >10% over the following 12 months; and,
* is not anticipated to need renal replacement therapy in the next 12 months; and,
* does not have any other clinical, biochemical or familial feature at screening that suggests a clinically significant decline in kidney function is anticipated in the next 12 months.

Exclusion Criteria:

For Part A:

* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study drug; or interfering with the interpretation of data.
* History of malignancy of any type.
* History of kidney disease or kidney abnormalities or eGFR less than (<) 90 milliliters per minute per 1.73 square meters (mL/min/1.73m^2) (based on the chronic kidney disease- Epidemiology Collaboration [CKD-EPI] 2021 eGFR equation) at screening.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study drug and for the duration of study participation.
* QT interval corrected (QTc)>450 milliseconds (msec)
* Participation in this study would result in loss of blood or blood products in excess of 500 mL within 56 days
* Current enrolment or past participation in an investigational clinical trial in which an investigational medicinal product was administered within the following time periods prior to the first dosing day of the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product, whichever is longer
* Exposure to more than 4 investigational medicinal products within 12 months prior to dosing
* Significant allergy to humanized monoclonal antibodies
* Clinically significant multiple or severe drug allergies, or severe post-treatment hypersensitivity reactions (including, but not limited to, erythema multiforme major, linear Immunoglobulin A (IgA) dermatosis, toxic epidermal necrolysis, and exfoliative dermatitis)
* Pregnant or lactating female
* Current or previous diagnosis of diabetes mellites (DM) (Type 1 or Type 2)
* Glycosylated hemoglobin (HbA1c) >=48 millimoles per mole (mmol/mol) (>=6.5%) at screening
* Bone fracture within 6 months prior to screening, or presence of a known unresolved or incompletely resolved fracture
* Positive pre-clinical study drug/alcohol screen, including tetrahydrocannabinol
* Positive Human Immunodeficiency Virus (HIV) antibody test
* Evidence of Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection, as determined by local diagnostic procedures
* Evidence at screening of clinically significant hematological disorder (affecting hemoglobin, red blood cells [RBC], White blood cells [WBC] or platelets) or abnormal blood clotting parameters
* Regular use of recreational drugs, including substances containing tetrahydrocannabinol
* Participants who are unable to refrain from smoking, vaping or using other tobacco products during study visits or overnight stays
* Poor peripheral venous access by visual inspection (intravenous [IV] administration cohort(s) only)
* Average weekly intake of greater than (>) 14 United Kingdom (UK) units of alcohol. One UK unit is equivalent to 8 grams (g) of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the investigator [or medical monitor], contraindicates participation in the study
* Use of any products intended to treat medical conditions that are not approved by the governing health authority in a given country or region (for example, herbal medicine, health supplements, traditional medicine, homeopathic remedies, etc.)
* Alanine transaminase (ALT) >1.5x Upper Limit of Normal (ULN)
* Total bilirubin >1.5xULN; Participants with Gilbert's syndrome can be included with total bilirubin <=3.0xULN as long as direct bilirubin is <=1.0xULN
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Presence of hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibody (HBcAb) at screening or within 3 months prior to first dose of study intervention
* Positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study intervention
* Positive hepatitis C Ribonucleic acid (RNA) test result at screening or within 3 months prior to first dose of study intervention

Part B:

* Presence of active, clinically significant cardiovascular, respiratory, hepatic, gastrointestinal, endocrine (including, but not limited to, incompletely controlled secondary or tertiary hyperparathyroidism and clinically significant vitamin D deficiency), hematological (including, but not limited to, transfusion-dependent anemia), bone (including, but not limited to, osteoporosis), or neurological disorders, with the exception of ADPKD, capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study drug; or interfering with the interpretation of data
* Clinically significant abnormal blood pressure (BP), that is, if the participant is not taking antihypertensive therapy: systolic BP >=160 millimeters of mercury (mmHg) and/or diastolic BP >=90mmHg; or If the participant is established on a stable regimen of antihypertensive drug(s): on-treatment systolic BP >=160 mmHg and/or diastolic BP >=90mmHg
* Lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of recurrence or metastatic disease for 3 years
* Breast cancer within the past 10 years
* Use of prescription and non-prescription drugs, including vitamins A, B, C, E, K, herbal and dietary supplements (including St John's Wort) within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study drug and for the duration of study participation. Paracetamol, at doses of <=4 gram per 24 hour (g/24h) is permitted for use at any time during the study
* Contraindication to, or unwillingness to undergo, MRI scanning (e.g., presence of MRI-incompatible metal implant)
* Congenital absence of one kidney
* Kidney cyst interventions such as cyst aspiration or cyst fenestration within 12 weeks prior to screening and during the screening period, or such interventions planned or anticipated within the follow-up period
* Acute symptomatic kidney cyst hemorrhage or infection within 12 weeks prior to screening
* Evidence of current, chronic, or recurrent kidney or liver cyst infection
* Estimated proteinuria >1g/24 hour at screening and/or pre-dose (day -7 to day -1)
* Abnormal urinalysis suggestive of clinically significant glomerular disease or urinary tract infection
* Presence of known clinically significant renal or hepatic calculi, or symptoms thereof, at screening
* Treatment with tolvaptan within 6 months prior to screening
* Presence of an incompletely healed wound at screening and/or planned surgical procedure that would occur during study.
* Participation in this study would result in loss of blood or blood products in excess of 500 mL within 56 days
* Current enrolment or past participation in an investigational clinical trial in which an investigational medicinal product was administered within the following time periods prior to the first dosing day of the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product, whichever is longer
* Exposure to more than 4 investigational medicinal products within 12 months prior to dosing
* Significant allergy to humanized monoclonal antibodies
* Clinically significant multiple or severe drug allergies, or severe post-treatment hypersensitivity reactions (including, but not limited to, erythema multiforme major, linear Immunoglobulin A (IgA) dermatosis, toxic epidermal necrolysis, and exfoliative dermatitis)
* Pregnant or lactating female
* Current or previous diagnosis of diabetes mellites (DM) (Type 1 or Type 2)
* HbA1c >=48 millimoles per mole (mmol/mol) (>=6.5%) at screening
* Bone fracture within 6 months prior to screening, or presence of a known unresolved or incompletely resolved fracture
* Positive pre-clinical study drug/alcohol screen, including tetrahydrocannabinol
* Positive HIV antibody test
* Evidence of SARS-CoV-2 infection, as determined by local diagnostic procedures
* Evidence at screening of clinically significant hematological disorder (affecting hemoglobin, RBC, WBC or platelets) or abnormal blood clotting parameters
* Regular use of recreational drugs, including substances containing tetrahydrocannabinol
* Participants who are unable to refrain from smoking, vaping or using other tobacco products during study visits or overnight stays
* Poor peripheral venous access by visual inspection (IV administration cohort(s) only)
* Average weekly intake of greater than (>) 14 UK units of alcohol. One UK unit is equivalent to 8 grams of alcohol: a half-pint (approximately240 mL) of beer, 1 glass (125 mL) of wine or 1 (25 mL) measure of spirits
* Sensitivity to any of the study interventions, or components thereof, or drug or other allergy that, in the opinion of the investigator [or medical monitor], contraindicates participation in the study
* Use of any products intended to treat medical conditions that are not approved by the governing health authority in a given country or region (for example, herbal medicine, health supplements, traditional medicine, homeopathic remedies, etc.)
* Alanine transaminase (ALT) >1.5x Upper Limit of Normal (ULN)
* Total bilirubin >1.5xULN; Participants with Gilbert's syndrome can be included with total bilirubin <=3.0xULN as long as direct bilirubin is <=1.0xULN
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Presence of HBsAg and/or HBcAb at screening or within 3 months prior to first dose of study intervention
* Positive hepatitis C antibody test result at screening or within 3 months prior to first dose of study intervention
* Positive hepatitis C RNA test result at screening or within 3 months prior to first dose of study intervention
* QTc >450 milliseconds (msec) or QTc >480 msec for participants with bundle branch block

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2026-09-04 (Estimated); Study Completion 2026-09-04 (Estimated)

PRIMARY OUTCOMES:
Part A: Number of Participants with Adverse events (AEs) | From Baseline (Day 1) up to Day 182 (End of study [EoS])
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention.
Part B: Number of Participants with AEs | From Baseline (Day 1) up to Day 182 (EoS)
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention.
Part A: Number of Participants with Serious Adverse Events (SAEs) | From Baseline (Day 1) up to Day 182 (EoS)
  An SAE is defined as any untoward medical occurrence that, at any dose, meets one or more of the criteria: results in death; is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant; abnormal pregnancy outcome (for example, spontaneous abortion, fetal death, stillbirth, congenital anomalies, ectopic pregnancy); is a suspected transmission of any infectious agent via an authorized medicinal product; or other situations.
Part B: Number of Participants with SAEs | From Baseline (Day 1) up to Day 182 (EoS)
  An SAE is defined as any untoward medical occurrence that, at any dose, meets one or more of the criteria: results in death; is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant; abnormal pregnancy outcome (for example, spontaneous abortion, fetal death, stillbirth, congenital anomalies, ectopic pregnancy); is a suspected transmission of any infectious agent via an authorized medicinal product; or other situations
Part A: Number of Participants with Clinically Significant Changes in Blood Laboratory Values | From Baseline (Day 1) up to Day 182 (EoS)
  Number of participants with clinically significant changes in blood laboratory values will be evaluated.
Part B: Number of Participants with Clinically Significant Changes in Blood Laboratory Values | From Baseline (Day 1) up to Day 182 (EoS)
  Number of participants with clinically significant changes in blood laboratory values will be evaluated.
Part A: Number of Participants with Clinically Significant Changes in Urine Laboratory Values | From Baseline (Day 1) up to Day 182 (EoS)
  Number of participants with clinically significant changes in Urine laboratory values will be evaluated.
Part B: Number of Participants with Clinically Significant Changes in Urine Laboratory Values | From Baseline (Day 1) up to Day 182 (EoS)
  Number of participants with clinically significant changes in Urine laboratory values will be evaluated.
Part A: Number of Participants with Clinically Significant Changes in Vital Signs | From Baseline (Day 1) up to Day 182 (EoS)
  Number of participants with clinically significant changes in vital signs (will be evaluated.
Part B: Number of Participants with Clinically Significant Changes in Vital Signs | From Baseline (Day 1) up to Day 182 (EoS)
  Number of participants with clinically significant changes in vital signs will be evaluated.
Part A: Number of Participants with Clinically Significant Changes in 12-lead Electrocardiogram (ECG) | From Baseline (Day 1) up to Day 182 (EoS)
  Number of participants with clinically significant changes in 12-lead ECG parameters will be evaluated.
Part B: Number of Participants with Clinically Significant Changes in 12-lead ECG | From Baseline (Day 1) up to Day 182 (EoS)
  Number of participants with clinically significant changes in 12-lead ECG parameters will be evaluated.

SECONDARY OUTCOMES:
Part A: Number of Participants with Anti-drug Antibodies for GSK4771261 | From Baseline (Day 1) up to Day 182 (EoS)
  Number of participants with Anti-drug antibodies for GSK4771261 will be evaluated.
Part B: Number of Participants with Anti-drug Antibodies for GSK4771261 | From Baseline (Day 1) up to Day 182 (EoS)
  Number of participants with Anti-drug antibodies for GSK4771261 will be evaluated.
Part A: Area under the concentration-time curve to the end of the dosing period AUC (0-tau) of GSK4771261 | Up to Day 182
  Blood samples were collected to evaluate pharmacokinetics of GSK4771261.
Part A: Area under the concentration-time curve to infinity AUC (0-inf) of GSK4771261 | Up to Day 182
  Blood samples were collected to evaluate pharmacokinetics of GSK4771261.
Part B: AUC (0-tau) of GSK4771261 | Up to Day 182
  Blood samples were collected to evaluate pharmacokinetics of GSK4771261.
Part B: AUC (0-inf) of GSK4771261 | Up to Day 182
  Blood samples were collected to evaluate pharmacokinetics of GSK4771261.
Part A: Maximum Plasma Concentration (Cmax) of GSK4771261 | Up to Day 182
  Blood samples were collected to evaluate of GSK4771261.
Part B: Cmax of GSK4771261 | Up to Day 182
  Blood samples were collected to evaluate of GSK4771261.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- Belgium (2):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Leuven
- Canada (2):
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Montreal, Quebec
- GSK Investigational Site, Brest, France
- GSK Investigational Site, Cologne, North Rhine-Westphalia, Germany
- Spain (2):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
- United Kingdom (4):
  - GSK Investigational Site, Cambridge
  - GSK Investigational Site, Exeter
  - GSK Investigational Site, London
  - GSK Investigational Site, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: Yes
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or asset(s) with development terminated across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months, but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/